CLINICAL TRIAL: NCT03561883
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Trial of Oral IW-3718 Administered to Patients With Gastroesophageal Reflux Disease While Receiving Proton Pump Inhibitors
Brief Title: Trial of IW-3718 for 8 Weeks in Patients With Persistent Gastroesophageal Reflux Disease (GERD) Receiving Proton Pump Inhibitors (PPIs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3718-302
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease; GERD; Proton Pump Inhibitor; IW-3718
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1500 mg IW-3718 BID (Experimental): Three 500 mg IW-3718 tablets administered twice daily (BID), immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
  Interventions: Drug: IW-3718; Drug: Standard-dose PPIs QD
- Placebo (Placebo Comparator): Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
  Interventions: Drug: placebo; Drug: Standard-dose PPIs QD

INTERVENTIONS:
Drug: IW-3718 — oral tablet
  Arms: 1500 mg IW-3718 BID
Drug: placebo — oral tablet
  Arms: Placebo
Drug: Standard-dose PPIs QD — background therapy

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of IW-3718 administered to patients with GERD who continue to have persistent symptoms, such as heartburn and regurgitation, while receiving once-daily (QD), standard dose PPIs.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be eligible for enrollment in this study:

* Patient is an ambulatory male or female (if female, nonpregnant) and is at least 18 years old at the Screening Visit.
* Patient has a diagnosis of GERD and reports experiencing GERD symptoms (heartburn or regurgitation) while taking standard PPI therapy.
* Patient has evidence of pathological acid reflux.
* Female patients must not be pregnant and must agree to avoid pregnancy for the duration of the study.
* Patient must comply with study procedures.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

* Patient has a history of complete lack of GERD symptom response to PPI therapy.
* Patient has a significant medical or surgical history including conditions that would impact drug absorption or metabolism (such as bowel obstruction, poorly controlled diabetes, gastroparesis, hiatal hernia).
* Patient reports pain or burning behind the breastbone or in the center of the upper stomach as his or her predominant symptom at the Screening Visit.
* Patient has received an investigational drug during the 30 days before the Screening Visit, or is planning to receive another investigational drug or use an investigational device at any time during the study.

NOTE: Other inclusion and exclusion criteria apply, per the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Shetzline, MD, PhD, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (99):
- United States (96):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialists of The Southeast, Dothan, Alabama
  - Holland Center for Family Health, Peoria, Arizona
  - Hope Research Institute LLC, Peoria, Arizona
  - Atria Clinical Research, Little Rock, Arkansas
  - Preferred Research Partners, Little Rock, Arkansas
  - Hope Clinical Research, LLC, Canoga Park, California
  - Om Research LLC, Lancaster, California
  - Torrance Clinical Research, Lomita, California
  - United Gastroenterologists, Murrieta, California
  - Clinical Applications Laboratories Inc, San Diego, California
  - Care Access Research, San Pablo, San Pablo, California
  - Paragon Rx Clinical, Inc. - Santa Ana, Santa Ana, California
  - Medical Research Center of Connecticut LLC, Hamden, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Optimus U Corp, Coral Gables, Florida
  - Nature Coast Clinical Research LLC - ERN-PPDS, Inverness, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Precision Clinical Research, LLC, Lauderdale Lakes, Florida
  - Suncoast Research Group LLC - ERN-PPDS, Miami, Florida
  - Applemed Research Inc, Miami, Florida
  - Gutierrez Medical Center, Orlando, Florida
  - Columbus Regional Research Institute at Talbotton, Columbus, Georgia
  - Consultative Gastroenterology, Decatur, Georgia
  - Atlanta Center For Clinical Research, Roswell, Georgia
  - Clinical Research Atlanta - ERN-PPDS, Stockbridge, Georgia
  - IL Gastroenterology Group, Gurnee, Illinois
  - Edward Hines Jr VA Hospital - NAVREF, Hines, Illinois
  - Aquiant Research, New Albany, Indiana
  - Kansas Medical Clinic, Topeka, Kansas
  - Heartland Research Associates LLC, Wichita, Kansas
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - Clinical Trials of America LA LLC, West Monroe, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Commonwealth Clinical Studies LLC, Brockton, Massachusetts
  - Center For Digestive Health, Troy, Michigan
  - Gastroenterology Associates of West Michigan, Wyoming, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - Gastrointestinal Associates PA, Flowood, Mississippi
  - Kansas City VA Medical Center - NAVREF, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Office of Michael Zimmerman, MD, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - NYScientific, Brooklyn, New York
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - United Health Services Hospitals, Johnson City, New York
  - Syracuse VA Medical Center - NAVREF, Syracuse, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Asheville Gastroenterology Associates PA, Asheville, North Carolina
  - UNC Medical Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Clinical Trials of America-NC, LLC, Mount Airy, North Carolina
  - PMG Research of Salisbury LLC, Salisbury, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - Hightop Medical Research Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - Dayton Gastroenterology Inc, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lynn Health Science Institute - ERN-PPDS, Oklahoma City, Oklahoma
  - Northwest Gastroenterology Clinic, Portland, Oregon
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Guthrie Research Institute, Sayre, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Trials of South Carolina - ClinEdge - PPDS, Charleston, South Carolina
  - Pharmacorp Clinical Trials Incorporated, Charleston, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Trials of South Carolina, North Charleston, South Carolina
  - Franklin Gastroenterology, Franklin, Tennessee
  - Clinical Research Solutions PC, Jackson, Tennessee
  - QUALITY Medical Research - Interspond - PPDS, Nashville, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Texas Health Physicians Group, Carrollton, Texas
  - Northside Gastroenterology, Cypress, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Coastal Medical Group, Houston, Texas
  - San Antonio Gastroenterology Associates Clinical Trials (SAGACT PLLC), San Antonio, Texas
  - Care Access Research, Salt Lake City, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Advanced Clinical Research - Gut Whisperer- ERN-PPDS, West Jordan, Utah
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - The Gastroenterology Group, Reston, Virginia
  - Clinical Research Partners LLC, Richmond, Virginia
  - Aurora Medical Center Summit, Summit, Wisconsin
  - Aurora Health Care, Waukesha, Wisconsin
- Canada (3):
  - Hughie Fraser, MD, Bridgewater, Nova Scotia
  - Viable Clinical Research, Bridgewater, Nova Scotia
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the screening and pre-treatment periods, participants were stratified by whether they had/did not have erosive esophagitis (EE) on esophagogastroduodenoscopy (EGD), and by their baseline weekly heartburn severity score (WHSS, defined as the average heartburn severity score over the last 7 days prior to randomization of < 3 vs. ≥ 3), and were randomly assigned 1:1 within each stratum to placebo or 1500 mg IW-3718 twice daily (BID).
Groups:
- Placebo BID + PPIs: Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose proton pump inhibitors (PPIs) administered once-daily (QD) approximately 30-60 minutes before the morning meal each day.
- 1500 mg IW-3718 BID + PPIs: Three 500 mg IW-3718 tablets administered BID, immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
Period: Overall Study
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs
Started | 305 | 304
Completed | 259 | 261
Not Completed | 46 | 43
Not completed — Adverse Event | 10 | 13
Not completed — Non-Compliance With Study Drug | 1 | 2
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 14 | 6
Not completed — Lost to Follow-up | 2 | 6
Not completed — Study Terminated by Sponsor | 12 | 11
Not completed — Physician Decision | 1 | 0
Not completed — Randomized by Mistake | 1 | 0
Not completed — Other, Not Specified | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: Participants who received at least 1 dose of study drug.
Groups:
- Placebo BID + PPIs: Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before the morning meal each day.
- Total: Total of all reporting groups
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs | Total
Number analyzed (Participants) | 304 | 304 | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.56) | 48.7 (12.61) | 49.3 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 187 | 373
  Male | 118 | 117 | 235
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 107 | 200
  Not Hispanic or Latino | 208 | 195 | 403
  Unknown | 3 | 0 | 3
  Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 233 | 246 | 479
  Black or African American | 63 | 49 | 112
  Asian | 3 | 5 | 8
  Other | 5 | 4 | 9
Erosive Esophagitis (EE) [Count of Participants; unit: Participants] — Population: Modified Intent-to-Treat (mITT) Population, which included all participants who 1) were randomized prior to or on 05 June 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
  Participants
    EE Present: number analyzed (Participants) | 276 | 277 | 553
    EE Present | 66 | 68 | 134
    EE Not Present: number analyzed (Participants) | 276 | 277 | 553
    EE Not Present | 210 | 209 | 419
Weekly Heartburn Severity Score (WHSS) Category [Count of Participants; unit: Participants] — WHSS=weekly average of Daily Heartburn Severity Score (DHSS). DHSS=the greater of the 2 items assessing heartburn severity (#1=Burning feeling behind the breastbone or in the center of the upper stomach; #2=Pain behind the breastbone or in the center of the upper stomach), where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms.
  Baseline is derived from the daily eDiary data collected in the pretreatment period, specifically the period of time from 7 days before randomization up to the time of randomization. Population: mITT Population, which included all participants who 1) were randomized prior to or on 05 June 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
  Participants
    WHSS Score ≥ 3: number analyzed (Participants) | 276 | 277 | 553
    WHSS Score ≥ 3 | 195 | 201 | 396
    WHSS Score < 3: number analyzed (Participants) | 276 | 277 | 553
    WHSS Score < 3 | 81 | 76 | 157
WHSS [Mean (Standard Deviation); unit: score on a scale] — WHSS=weekly average of DHSS. DHSS=the greater of the 2 items assessing heartburn severity (#1=Burning feeling behind the breastbone or in the center of the upper stomach; #2=Pain behind the breastbone or in the center of the upper stomach), where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms.
  Baseline is derived from the daily eDiary data collected in the pretreatment period, specifically the period of time from 7 days before randomization up to the time of randomization. Population: mITT Population, which included all participants who 1) were randomized prior to or on 05 June 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
  score on a scale
    number analyzed (Participants) | 276 | 277 | 553
    (all) | 3.32 (0.73) | 3.31 (0.72) | 3.32 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WHSS at Week 8
Description: The WHSS is defined as the weekly average of the DHSS. The DHSS for a day is the greater of the 2 items assessing heartburn severity (Item #1 "Burning feeling behind the breastbone or in the center of the upper stomach" and Item #2 "Pain behind the breastbone or in the center of the upper stomach"). The DHSS items are assessed on a 5-point ordinal scale, where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 8
Population: mITT Population: all participants who 1) were randomized prior to or on 05 June 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo BID + PPIs: Three placebo tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before morning meal each day.
- 1500 mg IW-3718 BID + PPIs: Three 500 mg IW-3718 tablets administered BID, immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before morning meal each day.
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs
Number analyzed (Participants) | 276 | 277
score on a scale | -1.751 (0.081) | -1.814 (0.082)
Statistical Analysis 1: Comparison: Placebo BID + PPIs vs 1500 mg IW-3718 BID + PPIs; Treatment difference calculated as least squares mean (LSM) change from baseline at Week 8; IW-3718 - placebo based on an mixed models repeated measures (MMRM) model with week (categorical), treatment group, week-by-treatment group and week-by-baseline value interactions, baseline esophagitis status (present vs. not present), and baseline WHSS (< 3 vs. ≥ 3) as fixed effect terms and baseline value as a covariate, with subject as a random effect. An unstructured covariance structure was used; Test type: Superiority; p = 0.5566, MMRM; Least squares (LS) mean difference = -0.062, 95% CI 2-sided [-0.270 to 0.146] — Treatment difference (IW-3718 - placebo)

2. Secondary Outcome: Change From Baseline in Weekly Regurgitation Frequency Score (WRFS) at Week 8
Description: The WRFS is defined as the average of available daily regurgitation frequency scores (DRFS) during a week. DRFS is defined as the maximum score of the 2 items measuring regurgitation from a particular day (Item #6 "Regurgitation [liquid or food moving upwards toward your throat or mouth]" and Item #7 "An acid or bitter taste in the mouth"). The DRFS items are assessed on a 4-point ordinal scale, where 0=Never, 1=Rarely, 2-Sometimes, 3=Often, and 4=Very Often; higher scores indicate worse symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs
Number analyzed (Participants) | 276 | 277
score on a scale | -1.278 (0.065) | -1.287 (0.065)
Statistical Analysis 1: Comparison: Placebo BID + PPIs vs 1500 mg IW-3718 BID + PPIs; Treatment difference calculated as LSM change from baseline at Week 8; IW-3718 - placebo based on an MMRM model with week (categorical), treatment group, week-by-treatment group and week-by-baseline value interactions, baseline esophagitis status (present vs. not present), and baseline WHSS (< 3 vs. ≥ 3) as fixed effect terms and baseline value as a covariate, with subject as a random effect. An unstructured covariance structure was used; Test type: Superiority; p = 0.9226, MMRM; LS mean difference = -0.008, 95% CI 2-sided [-0.176 to 0.159]

3. Secondary Outcome: Percentage of Participants Who Were Overall Heartburn Responders During the 8-Week Treatment Period
Description: An overall heartburn responder is a participant who is a weekly heartburn responder for at least 4 of the 8 treatment weeks and for at least 1 of the final 2 treatment weeks (i.e., Week 7 and Week 8). A weekly heartburn responder is a participant with a decrease of >/= 45% from baseline in WHSS. A participant who reported heartburn severity for less than 4 days during a week is not considered a responder for that week.
  The WHSS is defined as the weekly average of the DHSS. The DHSS for a day is the greater of the 2 items assessing heartburn severity (Item #1 "Burning feeling behind the breastbone or in the center of the upper stomach" and Item #2 "Pain behind the breastbone or in the center of the upper stomach"). The DHSS items are assessed on a 5-point ordinal scale, where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms. A negative change from baseline indicates improvement
Time Frame: Up to Week 8
Population: Modified Intent-to-Treat (mITT) Population: all participants who 1) were randomized prior to or on 05 June 2020, 2) had received at least 1 dose of study drug, and 3) had at least 1 postbaseline primary efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs
Number analyzed (Participants) | 276 | 277
percentage of participants | 41.3 | 42.6
Statistical Analysis 1: Comparison: Placebo BID + PPIs vs 1500 mg IW-3718 BID + PPIs; Test type: Superiority; Difference in Responder Rate = 1.3, 95% CI 2-sided [-6.9 to 9.5] — 95% confidence interval (CI) for Difference in Responder Rates is obtained using the Newcombe CI
Statistical Analysis 2: Comparison: Placebo BID + PPIs vs 1500 mg IW-3718 BID + PPIs; Treatment difference was calculated as the difference in the responder rates at Week 8; IW-3718 - placebo. The 95% CI for the difference in the responder rates was obtained using the Newcombe CI. P value was based on the odds ratio for the response rate (IW-3718:placebo) obtained from the Cochran-Mantel-Haenszel (CMH) tests controlling for baseline esophagitis status and baseline heartburn severity level (< 3 vs. ≥ 3); Test type: Superiority; p = 0.7424, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.76 to 1.48] — Odds Ratio for Response (IW-3718 : placebo)

4. Secondary Outcome: Proportion of Heartburn-Free Days During the 8-Week Treatment Period
Description: Proportion of heartburn-free days is calculated as the number of heartburn-free (DHSS=0) days divided by the number of diary entry days. The DHSS for a day is the greater of the 2 items assessing heartburn severity (Item #1 "Burning feeling behind the breastbone or in the center of the upper stomach" and Item #2 "Pain behind the breastbone or in the center of the upper stomach"). The DHSS items are assessed on a 5-point ordinal scale, where 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, and 5=Severe; higher scores indicate worse symptoms. A negative change from baseline indicates improvement
Time Frame: Up to Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: proportion of days
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs
Number analyzed (Participants) | 276 | 277
proportion of days | 0.200 (0.030) | 0.234 (0.033)
Statistical Analysis 1: Comparison: Placebo BID + PPIs vs 1500 mg IW-3718 BID + PPIs; Poisson regression including the fixed categorical effect of treatment, the baseline esophagitis status (present vs. not present) and baseline WHSS (<3 vs. ≥3), the covariate of baseline proportion of heartburn-free days, and with the diary entry duration (in days) as a weight variable adjusted in the model was applied; Test type: Superiority; p = 0.4164, Negative binomial model — Negative binomial model was used to deal with data overdispersion; Difference in Proportion Ratio = 1.171, 95% CI 2-sided [0.800 to 1.714] — Difference in Proportion Ratio, (1500 mg IW-3718 BID + PPI) - (Placebo + PPI)
Statistical Analysis 2: Comparison: Placebo BID + PPIs vs 1500 mg IW-3718 BID + PPIs; [analysis description as in outcome 4, analysis 1]; Test type: Other — Negative binomial model was used to deal with data overdispersion; Difference in Proportion Ratio = 0.034, 95% CI 2-sided [-0.054 to 0.123] — Difference in Proportion Ratio, (1500 mg IW-3718 BID + PPI) - (Placebo + PPI)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment (up to Week 8) plus 7 days.
Description: Safety Population: Participants who received at least 1 dose of study drug.
Groups:
- 1500 mg IW-3718 BID + PPIs: Three IW-3718 tablets administered BID immediately after the morning and evening meals. Standard-dose PPIs administered QD approximately 30-60 minutes before morning meal each day.
Arm/Group | Placebo BID + PPIs | 1500 mg IW-3718 BID + PPIs
All-Cause Mortality (participants affected / at risk) | 1/304 | 0/304
Serious Adverse Events (participants affected / at risk) | 3/304 | 2/304
Other Adverse Events (participants affected / at risk) | 6/304 | 15/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID + PPIs (N=304) | 1500 mg IW-3718 BID + PPIs (N=304)
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID + PPIs (N=304) | 1500 mg IW-3718 BID + PPIs (N=304)
Constipation (Gastrointestinal disorders) | 4 | 9
Nausea (Gastrointestinal disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03561883/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03561883/SAP_001.pdf